CLINICAL TRIAL: NCT03608033
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of the Safety and Efficacy of OMS721 in Patients With Immunoglobulin A (IgA) Nephropathy (ARTEMIS - IGAN)
Brief Title: Study of the Safety and Efficacy of OMS721 in Patients With Immunoglobulin A (IgA) Nephropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IA did not meet the prespecified primary endpoint.
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS721-IGA-001
Record Dates: First submitted 2018-06-21; First posted 2018-07-31 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; IgAN; Proteinuria; Chronic kidney disease; IgAN autoantibodies; eGFR; EGFR slope; UPE; Narsoplimab
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Renal Insufficiency, Chronic | interventions — narsoplimab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to receive OMS721 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OMS721 (Experimental): Administration of OMS721
  Interventions: Biological: OMS721
- Placebo (Placebo Comparator): Administration of Vehicle (D5W or Saline Solution)
  Interventions: Other: Vehicle (D5W or saline)

INTERVENTIONS:
Biological: OMS721 — Biological: OMS721
  Arms: OMS721
Other: Vehicle (D5W or saline) — 5% Dextrose in water or normal saline solution
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of OMS721 on 24-hour urine protein excretion (UPE) in IgA nephropathy (IgAN) patients with high baseline proteinuria (high-risk proteinuria group; 24-hour UPE ≥ 2 g/day) assessed at 36 weeks from baseline.

DETAILED DESCRIPTION:
This is a Phase 3, double-blind, randomized, placebo-controlled, study in patients aged 18 years and above with a biopsy-confirmed diagnosis of IgAN and with 24-hour UPE that is > 1 g/day. The purpose of this study is to evaluate the efficacy and safety of narsoplimab (OMS721) compared to placebo on proteinuria and whether narsoplimab has the ability to slow disease progression in primary IgAN patients. The primary objective of the study is to evaluate proteinuria reduction as assessed by 24-hour UPE at 36 weeks from baseline. The trial will continue beyond 36 weeks in a blinded fashion to provide confirmatory evidence of long-term efficacy based on the annualized slope of eGFR over 24 months. The trial will enroll approximately 450 patients with 225 patients per arm, all having biopsy-proven IgAN with eGFR≥30 mL/min/1.73m^2 and 24 hour UPE >1g/day. The study duration for each patient is expected to last approximately 112 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the onset of Screening
* Biopsy confirmed diagnosis of IgAN within 8 years prior to Screening or Run-in Visit 1
* Documented history of proteinuria of > 1 g/day within 6 months prior to Screening or uPCR > 0.75 by spot urine at Screening
* Mean of two proteinuria measurements > 1 g/day at baseline
* Estimated glomerular filtration rate of ≥ 30 mL/min/1.73 m² at Screening and baseline

Exclusion Criteria:

* Treatment with immunosuppressants (e.g., azathioprine or cyclophosphamide), Chinese traditional medicine with immunosuppressive function, cytotoxic drugs, or eculizumab within 8 weeks prior to Screening, unless such treatment is given for indications other than IgA.
* Treatment with systemic corticosteroids within 8 weeks prior to Screening
* Uncontrolled BP, a systolic BP of > 150 mmHg and a diastolic BP of > 100 mmHg at rest despite the combination of two or more anti-hypertensives including ACE inhibitors, ARBs, or direct renin inhibitors
* Female patients who are pregnant, breast feeding, or planning to become pregnant up through 12 weeks after the last dose of study drug, including possible retreatments. Males who are planning to father children up through 12 weeks after the last dose of study drug, including possible retreatments
* Clinical or biological evidence of Type 1 diabetes mellitus (DM), or poorly controlled DM with hemoglobin A1c > 7.5 or with evidence of diabetic nephropathy on biopsy, systemic lupus erythematosus, IgA vasculitis (Henoch-Schonlein purpura), secondary IgAN, or other renal disease during Screening and Run-In
* Presence of significant morbidity or other major illness or disease that may confound the interpretation of the clinical trial results or may result in death within 2 years of Screening
* History of renal transplantation
* Have a known hypersensitivity to any constituent of the investigational product
* Rapidly progressive glomerulonephritis, defined as a fall in eGFR of > 30 mL/min/1.73 m^2 within 24 weeks or > 15 mL/min/1.73 m^2 within 12 weeks prior to Screening
* Significant abnormalities in clinical laboratory values
* History of human immunodeficiency virus (HIV), evidence of immune suppression, active hepatitis C virus (HCV) infection (patients with positive anti-HCV antibody but a non-detected HCV RNA PCR can enroll), hepatitis B virus (HBV) infection (patients with positive HBsAg are excluded; for patients with isolated positive anti-HBc antibody, HBV DNA test by PCR must be non-detectable to enroll).
* Diagnosis of a malignancy except for adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or other cancer from which the patient has been disease-free for ≥ 5 years
* Have received any other investigational drug or device or experimental procedures within 30 days of the Screening Visit (SV) or within 5 times the plasma half-life of the administered experimental drug, whichever is longer
* Initiation or change in dosing of sodium glucose co-transporter 2 inhibitors (SGLT2i) during Screening and Run-In Periods. However, a stable dose regimen established at least 8 weeks prior to screening is acceptable
* Treatment with Tarpeyo™ (budesonide) or other approved treatments for IgAN within 6 months prior to screening. Treatment with Tarpeyo is not allowed during Screening and Run-In Periods
* Treatment with Kerendia® (finerenone) within 6 months prior to screening. Treatment with Kerendia is not allowed during Screening and Run-In Periods
* Initiation of treatment with Filspari™ (sparsentan), a dual Endothelin Angiotensin Receptor Antagonist (dEARA) or similar medication within three months prior to screening. A stable dose initiated at minimum 3 months before screening is acceptable and will take the place of ACEi/ARB as background therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (125):
- United States (32):
  - Omeros Investigational Site, Florence, Alabama
  - Omeros Investigational Site, Mesa, Arizona
  - Omeros Investigation Sites, Phoenix, Arizona
  - Omeros Investigational Site, Scottsdale, Arizona
  - Omeros Investigational Site, Los Angeles, California
  - Omeros Investigational Site, Northridge, California
  - Omeros Investigational Site, San Dimas, California
  - Omeros Investigational Site, San Francisco, California
  - Omeros Investigational Site, Stanford, California
  - Omeros Investigational Site, Torrance, California
  - Omeros Investigational Site, Denver, Colorado
  - Omeros Investigational Site, Miami, Florida
  - Omeros Investigational Site, Miami Lakes, Florida
  - Omeros Investigational Site, Lawrenceville, Georgia
  - Omeros Investigational Site, Chicago, Illinois
  - Omeros Investigational Site, Iowa City, Iowa
  - Omeros Investigational Site, Boston, Massachusetts
  - Omeros Investigational Site, Springfield, Massachusetts
  - Omeros Investigational Site, Minneapolis, Minnesota
  - Omeros Investigational Site, Rochester, Minnesota
  - Omeros Investigational Site, St Louis, Missouri
  - Omeros Investigational Site, Fresh Meadows, New York
  - Omeros Investigational Site, New York, New York
  - Omeros Investigational Site, Cincinnati, Ohio
  - Omeros Investigational Site, Columbus, Ohio
  - Omeros Investigational Site, Philadelphia, Pennsylvania
  - Omeros Investigational Site, Charleston, South Carolina
  - Omeros Investigational Site, Chattanooga, Tennessee
  - Omeros Investigational Site, Amarillo, Texas
  - Omeros Investigational Site, Dallas, Texas
  - Omeros Investigational Site, Houston, Texas
  - Omeros Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - Omeros Investigational Site, Posadas, Misiones Province
  - Omeros Investigational Site, Buenos Aires
  - Omeros Investigational Site, Córdoba
  - Omeros Investigational Site, Salta
- Australia (4):
  - Omeros Investigational Site, Garran, Australian Capital Territory, Woden
  - Omeros Investigational Site, Footscray, Saint Albans
  - Omeros Investigational Site, Adelaide, South Australia
  - Omeros Investigational Site, Clayton, Victoria
- Belgium (3):
  - Omeros Investigational Site, Ghent
  - Omeros Investigational Site, Leuven
  - Omeros Investigational Site, Liège
- Bulgaria (2):
  - Omeros Investigational Site, Plovdiv
  - Omeros Investigational Site, Sofia
- Canada (3):
  - Omeros Investigational Site, Vancouver, British Columbia
  - Omeros Investigational Site, London, Ontario
  - Omeros Investigational Site, Toronto, Ontario
- Omeros Investigational Site, Prague, Prague, Czechia
- Germany (5):
  - Omeros Investigational Site, Mannheim, Baden-Wrttemberg
  - Omeros Investigational Site, München, Bavaria
  - Omeros Investigational Site, Aachen, North Rhine-Westphalia
  - Omeros Investigational Site, Göttingen
  - Omeros Investigational Site, Villingen-Schwenningen
- Greece (4):
  - Omeros Investigational Site, Thessaloniki, Pilea-Chortiatis
  - Omeros Investigational Site, Athens
  - Omeros Investigational Site, Heraklion
  - Omeros Investigational Site, Pátrai
- Hungary (5):
  - Omeros Investigational Site, Baja
  - Omeros Investigational Site, Budapest
  - Omeros Investigational Site, Győr
  - Omeros Investigational Site, Pécs
  - Omeros Investigational Site, Szeged
- India (9):
  - Omeros Investigational Site, Hyderabad, Ameerpet
  - Omeros Investigational Site, Nadiād, Gujarat
  - Omeros Investigational Site, Belagavi, Karnataka
  - Omeros Investigational Site, Mangalore, Karnataka
  - Omeros Investigational Site, Kozhikode, Kerala
  - Omeros Investigational Site, New Delhi, New India
  - Omeros Investigational Site, Jaipur, Rajasthan
  - Omeros Investigational Site, Hyderabad, Telangana
  - Omeros Investigational Site, Chandigarh
- Italy (8):
  - Omeros Investigational Site, Bari
  - Omeros Investigational Site, Bergamo
  - Omeros Investigational Site, Eboli
  - Omeros Investigational Site, Messina
  - Omeros Investigational Site, Milan
  - Omeros Investigational Site, Modena
  - Omeros Investigational Site, Parma
  - Omeros Investigational Site, Piacenza
- Lithuania (2):
  - Omeros Investigational Site, Kaunas
  - Omeros Investigational Site, Vilnius
- Poland (4):
  - Omeros Investigational Site, Lodz, Todzi
  - Omeros Investigational Site, Krakow
  - Omeros Investigational Site, Olsztyn
  - Omeros Investigational Site, Warsaw
- Omeros Investigational Site, Singapore, Singapore
- Slovakia (2):
  - Omeros Investigational Site, Banská Bystrica
  - Omeros Investigational Site, Košice
- South Korea (5):
  - Omeros Investigational Site, Seongnam, Geyonggi-do
  - Omeros Investigational Site, Anyang-si, Gyeonggi-do
  - Omeros Investigational Site, Busan
  - Omeros Investigational Site, Incheon
  - Omeros Investigational Site, Seoul
- Spain (8):
  - Omeros Investigational Site, Madrid, San Sebastian de Lost Reyes
  - Omeros Investigational Site, Almería
  - Omeros Investigational Site, Barcelona
  - Omeros Investigational Site, Córdoba
  - Omeros Investigational Site, Lleida
  - Omeros Investigational Site, Madrid
  - Omeros Investigational Site, Valencia
  - Omeros Investigational Site, Zaragoza
- Omeros Investigational Site, Stockholm, Sweden
- Taiwan (6):
  - Omeros Investigational Site, Changhua
  - Omeros Investigational Site, Hualien City
  - Omeros Investigational Site, Kaohsiung City
  - Omeros Investigational Site, New Taipei City
  - Omeros Investigational Site, Taichung
  - Omeros Investigational Site, Taoyuan
- Thailand (5):
  - Omeros Investigational Site, Bangkok
  - Omeros Investigational Site, Chiang Mai
  - Omeros Investigational Site, Dusit
  - Omeros Investigational Site, Khon Kaen
  - Omeros Investigational Site, Songkhla
- Turkey (Türkiye) (6):
  - Omeros Investigational Site, Ankara
  - Omeros Investigational Site, Bursa
  - Omeros Investigational Site, Edirne
  - Omeros Investigational Site, Istanbul
  - Omeros Investigational Site, Kocaeli
  - Omeros Investigational Site, Malatya
- United Kingdom (5):
  - Omeros Investigational Site, Leicester, Evington
  - Omeros Investigational Site, Cambridge
  - Omeros Investigational Site, Cardiff
  - Omeros Investigational Site, Dartford
  - Omeros Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Karoui K, Fervenza FC, De Vriese AS. Treatment of IgA Nephropathy: A Rapidly Evolving Field. J Am Soc Nephrol. 2024 Jan 1;35(1):103-116. doi: 10.1681/ASN.0000000000000242. Epub 2023 Sep 29. PMID 37772889
- [Derived] Reich HN, Floege J. How I Treat IgA Nephropathy. Clin J Am Soc Nephrol. 2022 Aug;17(8):1243-1246. doi: 10.2215/CJN.02710322. Epub 2022 Jun 8. No abstract available. PMID 35675911

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with 24-hour UPE > 2 g/day at baseline will be allowed to receive 12-weeks of open-label active drug (OMS721) on Week 72 (18 months post randomization), provided they meet certain criteria:
  * Less than 30% reduction in UPE at the OL assessment visit from baseline UPE
  * Proteinuria is ≥ 3.0 g/day at 72 weeks from randomization, confirmed by 2 measurements at least 2 weeks apart, but < 3 weeks
  * Worsening renal function, defined as a decline in eGFR of > 5 mL/min/m^2 from baseline
Period: Treatment Period
Arm/Group | OMS721 | Placebo
Started | 181 | 179
Completed | 37 | 39
Not Completed | 144 | 140
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 5
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 2 | 6
Not completed — Physician Decision | 6 | 10
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 46 | 45
Not completed — Study terminated by sponsor | 82 | 68
Not completed — Site Terminated by Sponsor | 1 | 0
Period: Open-Label Period: OMS721
Arm/Group | OMS721 | Placebo
Started | 34 | 0
Completed | 15 | 0
Not Completed | 19 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Terminated By Sponsor | 11 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMS721 | Placebo | Total
Number analyzed (Participants) | 181 | 179 | 360
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 40.7 (12.01) | 41.6 (12.76) | 41.2 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 61 | 128
  Male | 114 | 118 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 11 | 33
  Not Hispanic or Latino | 157 | 166 | 323
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 52 | 62 | 114
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 120 | 112 | 232
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Child Bearing Potential, n (%) [Number; unit: participants]
  Yes | 49 | 45 | 94
  No | 18 | 16 | 34
  Not Applicable (Male Subjects) | 114 | 118 | 232
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: Two participants were treated with OMS721 without following appropriate randomization procedures resulting in major protocol deviations. Thus, these participants were not included in the analysis population. One participant in the placebo group was randomized but did not have weight collected.
  kg
    number analyzed (Participants) | 179 | 178 | 357
    (all) | 82.7 (19.95) | 82.5 (22.39) | 82.6 (21.17)
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] — Population: Two participants were treated with OMS721 without appropriate randomization procedures resulting in major protocol deviations. Thus, these participants were not included in this analysis. One subject in the placebo group was randomized but did not have height collected.
  cm
    number analyzed (Participants) | 179 | 178 | 357
    (all) | 170.8 (9.39) | 171.9 (10.10) | 171.4 (9.75)
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  kg/m^2
    number analyzed (Participants) | 179 | 179 | 358
    (all) | 28.3 (6.51) | 27.8 (6.87) | 28.1 (6.69)
Baseline Systolic Blood Pressure (mmHG) [Mean (Standard Deviation); unit: mmHg] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  mmHg
    number analyzed (Participants) | 179 | 179 | 358
    (all) | 125.7 (10.13) | 124.8 (12.03) | 125.3 (11.11)
Baseline Diastolic Blood Pressure (mmHG) [Mean (Standard Deviation); unit: mmHg] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  mmHg
    number analyzed (Participants) | 179 | 179 | 358
    (all) | 78.3 (8.3) | 77.8 (9.15) | 78.1 (8.72)
Baseline Estimated Glomerular Filtration Rate (mL/min/SSA), n(%) [Number; unit: participants] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  participants
    Greater than or equal to 30 and Less than or equal to 45: number analyzed (Participants) | 179 | 179 | 358
    Greater than or equal to 30 and Less than or equal to 45 | 63 | 62 | 125
    Greater than 45: number analyzed (Participants) | 179 | 179 | 358
    Greater than 45 | 116 | 117 | 233
Baseline Urine Protein Excretion Rate (mg/24hrs) [Mean (Standard Deviation); unit: mg/24hrs] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  mg/24hrs
    number analyzed (Participants) | 179 | 179 | 358
    (all) | 2780.5 (1633.49) | 2869.3 (1802) | 2824.9 (1717.98)
Baseline Urine Protein Creatinine Ratio [Mean (Standard Deviation); unit: (g/g)] — Population: Two patients were not randomized correctly in accordance with protocol procedures resulting in major protocol deviations. The patients were assigned to a treatment arm before study drug was administered. Therefore, these participants were not included in this analysis.
  (g/g)
    number analyzed (Participants) | 179 | 179 | 358
    (all) | 2.0 (1.21) | 2.1 (1.19) | 2.1 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in 24-hour UPE in g/Day Compared to Baseline
Description: The Primary Endpoint of this Study is the Percent Change from Baseline in Log-transformed 24-hour UPE in g/Day at 36 Weeks in Patients with High Baseline Proteinuria (High-risk Proteinuria Group; 24-hour UPE ≥ 2 g/day.
Time Frame: 36 Weeks
Population: The prespecified Primary Interim Analysis was in patients who had a 24-hour UPE ≥ 2 g/day at baseline. The study was terminated after the Primary Analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 70 | 69
Percent Change | -21.3 (0.0672) | -16.6 (0.0680)

2. Secondary Outcome: Change in Annualized eGFR Compared to Baseline.
Description: The Rate of Change in eGFR up to 96 Weeks from Baseline in Patients with High Baseline Proteinuria (High-risk Proteinuria Group; 24-hour UPE ≥ 2 g/Day)
Time Frame: 96 Weeks
Population: The prespecified secondary outcome analysis was in patients who had a 24-hour UPE ≥ 2 g/day at baseline. Since the study was terminated early, not all patients reached week 96, therefore the last observation was carried forward for analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²/year
Groups:
- OMS721 (High Baseline Proteinuria Group): High-risk Proteinuria Patients; 24-hour UPE ≥ 2 g/Day
  Biological: OMS721
- Placebo (High Baseline Proteinuria Group): High-risk Proteinuria Patients; 24-hour UPE ≥ 2 g/Day
  Placebo
Arm/Group | OMS721 (High Baseline Proteinuria Group) | Placebo (High Baseline Proteinuria Group)
Number analyzed (Participants) | 112 | 111
mL/min/1.73 m²/year | -8.3 (0.9) | -7.9 (0.9)

3. Secondary Outcome: Change in Annualized eGFR Compared to Baseline in All Patients.
Description: The Rate of Change in eGFR up to 96 Weeks from Baseline in the All-patients Population (24-hour UPE > 1 g/Day)
Time Frame: 96 Weeks
Population: The prespecified secondary outcome analysis was in patients who had a 24-hour UPE > 1 g/day at baseline. Since the study was terminated early, not all patients reached week 96, therefore the last observation was carried forward for analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²/year
Groups:
- Placebo: Administration of Placebo
  Placebo
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 179 | 178
mL/min/1.73 m²/year | -6.4 (0.7) | -7.6 (0.7)

4. Secondary Outcome: Change in 24-hour UPE in g/Day Compared to Baseline in All Patients
Description: Change From Baseline in Log-transformed 24-hour UPE at Week 36 in the All-patients Population. (24-hour UPE > 1 g/Day)
Time Frame: 36 Weeks
Population: Outcome data for this secondary outcome measure are available for a subset of 260 of the 360 participants (132 OMS721 and 128 placebo). These data are presented. Because the data collected up to the time of study termination for this outcome measure are incomplete, reliance on these measures could provide inaccurate and/or misleading information.
Measure: Mean (Standard Deviation); unit: g/ 24hrs
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 132 | 128
g/ 24hrs | -14.2 (0.7) | -10.3 (0.6)

5. Secondary Outcome: Change in 24-hour UPE in g/Day Between 36 Weeks and 48 Weeks.
Description: Change From Baseline in the Log-transformed 24-hour UPE Between 36 Weeks and 48 Weeks in Patients With ≥ 2 g/Day UPE at Baseline (High-risk Proteinuria Group)
Time Frame: 36 weeks and 48 weeks
Population: Outcome measure data for this secondary outcome measure are available for a subset of 131 of the 180 participants (66 OMS721 and 65 placebo). These data are presented. Because the data collected up to the time of study termination for this outcome measure are incomplete, reliance on the data could provide inaccurate and/or misleading information.
Measure: Mean (Standard Deviation); unit: g/24hr
Groups:
- OMS721 (High-risk Proteinuria Group): Patients With ≥ 2 g/Day UPE at Baseline (High-risk Proteinuria Group)
  Administration of OMS721
  OMS721: Biological: OMS721
- Placebo (High-risk Proteinuria Group): Patients With ≥ 2 g/Day UPE at Baseline (High-risk Proteinuria Group)
  Administration of Vehicle (D5W or Saline Solution)
  Vehicle (D5W or saline): 5% Dextrose in water or normal saline solution
Arm/Group | OMS721 (High-risk Proteinuria Group) | Placebo (High-risk Proteinuria Group)
Number analyzed (Participants) | 66 | 65
g/24hr | 4.1 (0.5) | 4.4 (0.6)

6. Secondary Outcome: Change in 24-hour UPE in g/Day Between 36 Weeks and 72 Weeks in Patients With >= 2 g/Day UPE at Baseline (High-risk Proteinuria Group).
Description: Time-averaged Change from Baseline in the Log-transformed 24-hour UPE Between 36 Weeks and 72 Weeks in Patients with ≥ 2 g/Day UPE at Baseline (High-risk Proteinuria Group)
Time Frame: 36 weeks and 72 weeks
Population: Outcome measure data for this secondary outcome measure are available for a subset of 121 of the 180 participants (60 OMS721 and 61 placebo). These data are presented. Because the data collected up to the time of study termination for this outcome measure are incomplete, reliance on the data could provide inaccurate and/or misleading information.
Measure: Mean (Standard Deviation); unit: g/24hr
Arm/Group | OMS721 (High-risk Proteinuria Group) | Placebo (High-risk Proteinuria Group)
Number analyzed (Participants) | 60 | 61
g/24hr | 11.6 (0.7) | 7.5 (0.8)

7. Secondary Outcome: Change in 24-hour UPE in g/Day Between 36 Weeks and 48 Weeks in All Patients
Description: Time-averaged Change from Baseline in the Log-transformed 24-hour UPE Between 36 Weeks and 48 Weeks in the All-patients Population
Time Frame: 36 weeks and 48 weeks
Population: Outcome measure data for this secondary outcome measure are available for a subset of 229 of the 360 participants (118 OMS721 and 111 placebo). These data are presented. Because the data collected up to the time of study termination for this outcome measure are incomplete, reliance on the data could provide inaccurate and/or misleading information.
Measure: Mean (Standard Deviation); unit: g/24hr
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 118 | 111
g/24hr | 6.2 (0.5) | 3.5 (0.6)

8. Secondary Outcome: Change in 24-hour UPE in g/Day Between 36 Weeks and 72 Weeks in All Patients
Description: Time-averaged Change from Baseline in the Log-transformed 24-hour UPE between 36 Weeks and 72 Weeks in the All-patients Population
Time Frame: 36 weeks and 72 weeks
Population: Outcome measure data for this secondary outcome measure are available for a subset of 203 of the 360 participants (103 OMS721 and 100 placebo). These data are presented. Because the data collected up to the time of study termination for this outcome measure are incomplete, reliance on the data could provide inaccurate and/or misleading information.
Measure: Mean (Standard Deviation); unit: g/24hr
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 103 | 100
g/24hr | 10.9 (0.7) | 14.2 (0.8)

9. Secondary Outcome: Safety and Tolerability of Narsoplimab for the Treatment of IgAN as Assessed by AEs, Vital Signs, Clinical Laboratory Tests, and ECGs
Description: As assessed by the incidence of adverse events through study completion (Week 112) in the patient group in the all-patients population. Clinically meaningful abnormalities in vital signs, clinical laboratory tests, and ECGs were collected as AEs.
Time Frame: Week 112
Population: Any patient who received study drug (N=360)
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 | Placebo
Number analyzed (Participants) | 181 | 179
Participants | 181 | 179

ADVERSE EVENTS:
Time Frame: The Adverse Event period of time was from the date of Consent to up to 112 weeks (includes Screen and Run-in) or end of study visit
Description: Treatment-emergent AEs are assessed throughout the study from first dose up to 96 weeks or end of study visit. Treatment-emergent AEs during blinded phase are displayed separately from Open-label phase.
Groups:
- Open-Label OMS721: Subgroup of patients from blinded (either treatment group) who subsequently received open-label OMS721 during the open-label period
  OMS721: Biological: OMS721
Arm/Group | OMS721 | Placebo | Open-Label OMS721
All-Cause Mortality (participants affected / at risk) | 0/181 | 1/179 | 0/34
Serious Adverse Events (participants affected / at risk) | 22/181 | 20/179 | 7/34
Other Adverse Events (participants affected / at risk) | 137/181 | 121/179 | 25/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMS721 (N=181) | Placebo (N=179) | Open-Label OMS721 (N=34)
SAE by System Organ (Infections and infestations) | 7 | 7 | 3
SAE by System Organ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
SAE by System Organ (Blood and lymphatic system disorders) | 1 | 2 | 0
SAE by System Organ (Immune system disorders) | 1 | 1 | 0
SAE by System Organ (Metabolism and nutrition disorders) | 2 | 3 | 0
SAE by System Organ (Nervous system disorders) | 2 | 0 | 0
SAE by System Organ (Ear and labyrinth disorders) | 0 | 1 | 0
SAE by System Organ (Cardiac disorders) | 0 | 2 | 0
SAE by System Organ (Vascular disorders) | 1 | 0 | 0
SAE by System Organ (Gastrointestinal disorders) | 3 | 0 | 1
SAE by System Organ (Hepatobiliary disorders) | 1 | 0 | 0
SAE by System Organ (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
SAE by System Organ (Renal and urinary disorders) | 9 | 7 | 4
SAE by System Organ (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
SAE by System Organ (General disorders) | 1 | 2 | 0
SAE by System Organ (Injury, poisoning and procedural complications) | 1 | 3 | 0
SAE by System Organ (Product Issues) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMS721 (N=181) | Placebo (N=179) | Open-Label OMS721 (N=34)
AE by System Organ (Blood and lymphatic system disorders) | 13 | 9 | 2
AE by System Organ (Cardiac disorders) | 8 | 5 | 2
AE by System Organ (Congenital, familial and genetic disorders) | 0 | 2 | 0
AE by System Organ (Endocrine disorders) | 5 | 3 | 1
AE by System Organ (Eye disorders) | 9 | 3 | 1
AE by System Organ (Gastrointestinal disorders) | 42 | 38 | 4
AE by System Organ (General disorders) | 49 | 34 | 8
AE by System Organ (Hepatobiliary disorders) | 4 | 0 | 8
AE by System Organ (Immune system disorders) | 3 | 2 | 0
AE by System Organ (Infections and infestations) | 89 | 73 | 14
AE by System Organ (Injury, poisoning and procedural complications) | 22 | 16 | 2
AE by System Organ (Investigations) | 24 | 17 | 7
AE by System Organ (Metabolism and nutrition disorders) | 29 | 18 | 3
AE by System Organ (Musculoskeletal and connective tissue disorders) | 40 | 26 | 8
AE by System Organ (Nervous system disorders) | 33 | 36 | 2
AE by System Organ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0
AE by System Organ (Product Issues) | 1 | 0 | 0
AE by System Organ (Psychiatric disorders) | 5 | 6 | 1
AE by System Organ (Renal and urinary disorders) | 28 | 24 | 5
AE by System Organ (Reproductive system and breast disorders) | 10 | 5 | 1
AE by System Organ (Respiratory, thoracic and mediastinal disorders) | 28 | 15 | 3
AE by System Organ (Skin and subcutaneous tissue disorders) | 22 | 23 | 3
AE by System Organ (Surgical and medical procedures) | 1 | 0 | 0
AE by System Organ (Vascular disorders) | 20 | 19 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs are restricted from publishing the results of the study until after sponsor publishes or 18 months after end of study at all sites. Sponsor requires removal of confidential information

DOCUMENTS (2):
  • Study Protocol (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03608033/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03608033/SAP_001.pdf